CLINICAL TRIAL: NCT03808363
Title: High-intensity Interval Training Versus Moderate Intensity Continuous Training as a Means to Improve Cardiometabolic Health After Spinal Cord Injury
Brief Title: Effectiveness of High Intensity Interval Training (HIIT) on Improving Cardiometabolic Health After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, David Ditor, David Ditor, PhD - Professor, Kinesiology, Brock University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-022-DITOR
Record Dates: First submitted 2018-10-22; First posted 2019-01-17 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Metabolic Syndrome; Cardiovascular Diseases
Keywords: Metabolic Syndrome; Spinal Cord Injury; Cardiovascular Disease; High Intensity Interval Training
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Spinal Cord Injuries | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 6 week exercise intervention testing the efficacy of high intensity interval training as compared to current research supporting moderate intensity continuous exercise as a means to mitigate cardiometabolic decline following spinal cord injury
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Interval Training Group (Experimental): Approximately eight individuals with spinal cord injuries will participate in high intensity interval training for 6 weeks
  Interventions: Other: High Intensity Interval Training

INTERVENTIONS:
Other: High Intensity Interval Training — Participants assigned to this group will perform a very mild 5-minute warm-up (0 resistance, and 60 rpm), followed by 5 one-minute bouts of high intensity exercise, with 90 seconds between each bout. These bouts will be followed by a 3-minute cool down (0 resistance, and 60 rpm). The high-intensity exercise will be performed at an intensity of 17 on the Borg rating of perceived exertion (RPE) scale (very hard), and the 90 second active rest intervals will be performed at an intensity of 7-9 (very, very light - very light). The exercise will be performed on the NuStep machine 3 times a week for 6 weeks.
  Other Names: HIIT

SUMMARY:
Testing the efficacy of high intensity interval training (HIIT), as compared to current research supporting moderate intensity continuous training (MICT), as a means to improve cardiometabolic health after spinal cord injury.

DETAILED DESCRIPTION:
This study aims to challenge the effectiveness of the current aerobic exercise recommendations for individuals with spinal cord injuries (SCI). Currently, moderate intensity continuous training (MICT) is suggested however this study intends to explore the effectiveness of high intensity interval training (HIIT). To do so, approximately 8 individuals with SCI will be undergo a 6 week HIIT intervention consisting of 3 sessions per week. With a focus on cardiometabolic health markers (listed in outcome measure section), we aim to provide support for HIIT as a viable method of mitigating cardiovascular risk in a SCI population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a spinal cord injury (paraplegia or tetraplegia, complete or incomplete) who are at least one-year post injury.
* Declared medically stable, and able to communicate clearly in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Waist circumference (inches) | 6 weeks
  Central adiposity will be measured by tape measure to monitor possible weight loss
Cholesterol | 6 weeks
  Total and HDL cholesterol will be measured in serum
Triglycerides | 6 weeks
  Triglycerides will be measured in serum
Glycated Hemoglobin (HbA1c) | 6 weeks
  Glycated hemoglobin will be measured in whole blood as an indicator of diabetic risk
Tumor necrosis factor (TNF-a) | 6 weeks
  TNF-a will be used as an inflammatory representative and will be measured in serum
Interleukin - 10 (IL-10) | 6 weeks
  IL-10 will will be used as an anti-inflammatory representative and will be measured in serum
Pulse Wave Velocity | 6 weeks
  Arterial stiffness, a common measure for cardiac risk will be measured
Blood pressure | 6 weeks
  Measured through a digital cuff, the focus will be on both systolic and diastolic
Peak Oxygen Consumption (VO2 peak) | 6 weeks
  VO2 peak will be measured by a Moxus metabolic cart to determine changes in fitness
C Reactive Protein (CRP) | 6 weeks
  CRP will will be used as an inflammatory representative and will be measured in serum
Leptin | 6 weeks
  Leptin will will be used as a body fat representative and will be measured in serum
Adiponectin | 6 weeks
  Adiponectin will will be used as a surrogate for insulin resistance and will be measured in serum

SECONDARY OUTCOMES:
Physical Activity Enjoyment Scale (PACES) | 6 weeks
  All participants will complete the physical activity enjoyment scale (PACES) to indicate enjoyment of HIIT. With a total of 18 questions, options 1 through 7 going from a positive to a negative overall experience with the HIIT protocol will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel Gibson, BKin, Principal Investigator — Masters Student; Aaron Donst, BKin, Principal Investigator — Masters Student
Locations (1):
- Brock University, Saint Catherines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No